CLINICAL TRIAL: NCT00971399
Title: Phase III Prospective Randomized Trial Comparing Ramosetron Versus Ondansetron for Radiotherapy Induced Nausea and Vomiting in the Treatment of Gastrointestinal Cancer
Brief Title: Ramosetron Versus Ondansetron for Radiotherapy Induced Nausea and Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Eui Kyu Chie/Assistant Clinical Professor, Department of Radiation Oncology, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RMS vs ODS for CRINV; 0808-011-252
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Radiotherapy Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — ramosetron; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RMS (Experimental): ramosetron 0.1mg q.d. SL on D1-5
  Interventions: Drug: ramosetron
- ODS (Active Comparator): ondansetron 8mg, b.i.d SL on D1-5
  Interventions: Drug: ondansetron

INTERVENTIONS:
Drug: ramosetron — ramosetron 0.1mg q.d. SL on D1-5
  Arms: RMS
Drug: ondansetron — ondansetron 8mg, b.i.d SL on D1-5
  Arms: ODS

SUMMARY:
The purpose of this study is:

1. To compare prophylactic effect of ondansetron versus ramosetron on radiotherapy induced nausea and vomiting in the treatment of gastrointestinal cancer.
2. To verify an improvement of 20% in complete response rate in term of radiotherapy induced nausea and vomiting (from 60% with ondansetron to 80% with ramosetron).

ELIGIBILITY:
Inclusion Criteria:

* AJCC 1-3 staged gastrointestinal cancer patient
* patient undergoing radiotherapy as treatment
* age 20 yr and higher
* ECOG 0-2

Exclusion Criteria:

* age < 20
* ECOG 3-4
* patient experiencing nausea or vomiting prior to accrual
* patient under antiemetic medication
* patient under steroid medication (topical or inhalant steroid application are exceptional)
* patient under opioid medication

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
complete response of RINV (no vomiting and no rescue medication) | 4 weeks after medication

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Kim K, Chie EK, Jang JY, Kim SW, Oh DY, Im SA, Kim TY, Bang YJ, Ha SW. Ramosetron for the prevention of nausea and vomiting during 5-fluorouracil-based chemoradiotherapy for pancreatico-biliary cancer. Jpn J Clin Oncol. 2009 Feb;39(2):111-5. doi: 10.1093/jjco/hyn140. Epub 2008 Dec 5. PMID 19060294